CLINICAL TRIAL: NCT01834508
Title: A 3-year, Open-lable, Multi-center Extension Trial of Entecavir Plus Adefovir Combination Treatment for Patients Previously Treated in EXPLORE, EXCEL and EFFORT Ex Study
Brief Title: 3E Extension Study
Acronym: 3E Ex
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Collaborators: Major Science and Technology Special Project of China 12th Five-year (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MOH-07
Record Dates: First submitted 2013-04-14; First posted 2013-04-18 (Estimated); Last update posted 2014-06-19 (Estimated); Status verified 2014-06

CONDITIONS: Chronic Hepatitis B
Keywords: Experienced Treatment
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — entecavir; adefovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment group (Other)
  Interventions: Drug: oral entecavir 0.5mg daily and adefovir 10mg daily for 144 weeks

INTERVENTIONS:
Drug: oral entecavir 0.5mg daily and adefovir 10mg daily for 144 weeks

SUMMARY:
The purpose of this study is to evaluate the long-term efficacy and safety of entecavir 0.5 mg/d + adefovir 10 mg/d for treatment experienced chronic hepatitis B patients.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who completed the EXPLORE or EXCEL studies, or subjects with hepatitis flare after treatment withdrawal in EFFORT study.
* Subjects who are willing to participate the extension study.

Exclusion Criteria:

* Subjects who could not compliance with the protocol judged by investigators

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2013-03; Primary Completion 2016-06 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Percentages of patients achieving HBV DNA< 300copies/mL at week 144 | Week 144

SECONDARY OUTCOMES:
Percentages of patients achieving HBV DNA <300copies/mL at week 48/96 | Week 48 & 96
The log10 reduction in HBV DNA from baseline of DRAGON study at week 48/96/144 | Week 48 & 96 &144
Percentage of patients with HBeAg loss or HBeAg seroconversion at week 48/96/144. | Week 48 & 96 & 144
Percentage of patients with ALT normalization at week 48/96/144 | Week 48 & 96 & 144

CONTACTS AND LOCATIONS:
Locations (28):
- China (28):
  - 302 Military Hospital Of China, Beijing, Beijing Municipality
  - Beijing Ditan Hospita, Beijing, Beijing Municipality
  - Beijing Friendship Hospital Attached To The Capital Medical University, Beijing, Beijing Municipality
  - BeiJing YouAn Hospital ,Capital Medical University, Beijing, Beijing Municipality
  - Department of infectious disease, First Hospital of Peking University, Beijing, Beijing Municipality
  - People's Hospital Under Beijnig University, Beijing, Beijing Municipality
  - The Second Affiliated of ChongQing University of Medical Science, Chongqing, Chongqing Municipality
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian
  - The First People's Hospital of Foshan, Foshan, Guangdong
  - Department of Infectious Disease, Nanfang Hospital, Guangzhou, Guangdong
  - GuangDong Provincial People's hospital, Guangzhou, Guangdong
  - No. 8 People's Hospital In GuangZhou, Guangzhou, Guangdong
  - The Third Hospital of Sun Yat-Sen University, Guangzhou, Guangdong
  - First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi
  - Tongji Hospital of Tongji Medical College of Huazhong University of Science and Technology, Wuhan, Hubei
  - Xiangya Hospital Central-South Univrsity, Changsha, Hunan
  - No.81 Hospital of PLA, Nanjing, Jiangsu
  - First Hospital .Jilin Unniversity, Changchun, Jilin
  - ShengJing Hospital of China Medical University, Shengyang, Liaoning
  - JiNan Infectious Diseases Hospital, Jinan, Shandong
  - Changhai Hospital affiliated to Second Military Medical University, Shanghai, Shanghai Municipality
  - Huashan Hospital，Fudan University, Shanghai, Shanghai Municipality
  - No.85 Hospital of PLA, Shanghai, Shanghai Municipality
  - Shanghai Ruijin Hospital, Shanghai, Shanghai Municipality
  - Tangdu Hospital, XiAn, Shanxi
  - West China Hospital.SiChuan University, Chengdu, Sichuan
  - HangZhou No.6 People Hospital, Hangzhou, Zhejiang
  - The First Affiliated Hospital of College of Medicine, Zhejiang University, Hangzhou, Zhejiang